CLINICAL TRIAL: NCT02839174
Title: Investigation of Glycemic Control Among an International Community of People With Type 1 Diabetes Following a Low Carbohydrate Diet
Brief Title: Type One Diabetes and Low Carb Study
Status: Completed | Type: Observational
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Belinda Lennerz, Instructor in Pediatric Endocrinology, Boston Children's Hospital
Other Study IDs: P00022864
Record Dates: First submitted 2016-07-14; First posted 2016-07-20 (Estimated); Last update posted 2017-06-09 (Actual); Status verified 2017-06

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: low carbohydrate diet
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
The investigators have identified a support group on social media with ~1500 members (children and adults), the majority of whom have T1DM and follow a carbohydrate-restricted diet. Many participants report exceptionally low HbA1C and insulin requirements. If these anecdotal reports are reflective of a large group of people with type 1 diabetes, a clinical trial would be warranted.

The investigators propose to survey the above-mentioned group and their professional diabetes care providers to characterize glycemic control and explore associated dietary and diabetes care factors.

DETAILED DESCRIPTION:
The surveys will address questions in the following domains: 1) Diabetes diagnosis and treatment; 2) Carbohydrate-restricted diet; 3) Insulin regimen; 4) Other diabetes related care; 5) Diabetes complications; 6) Other related health and healthcare; 7) Patient provider interactions; 8) Socio-demographics. Drafts of these surveys are included in the appendix of this protocol.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with a diagnosis of T1DM who are currently on insulin treatment or
* Adults who are a parent or guardian of a child with T1DM who is currently on insulin treatment and
* Self-reported use of a regimen including carbohydrate restriction for at least 3 months

Exclusion Criteria:

* Women who are pregnant or breastfeeding.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The social media group on Facebook, TYPEONEGRIT, includes approximately 1500 members, the majority of whom reportedly have type 1 diabetes and follow a carbohydrate-restricted diet.
Sampling Method: Non-Probability Sample
Enrollment: 340 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Hemoglobin A1C | within 3 month of taking the survey
  self reported, confirmed by professional diabetes care provider if possible

SECONDARY OUTCOMES:
total daily insulin dose | within 3 month of taking the survey
  self reported, confirmed by professional diabetes care provider if possible
total daily dietary carbohydrate | within 3 month of taking the survey
  self reported
diabetes-related complication rates - diabetic ketoacidosis, hypoglycemia | timeframe since staring low carb diet (at least three months)
BMI | within 3 month of taking the survey
  self reported, confirmed by professional diabetes care provider if possible
change in HbA1C | current (within three months of taking the survey) - baseline (last available pre-carbohydrate-restricted diet)
  self reported, confirmed by professional diabetes care provider if possible
patient-physician relationship | within 3 month of taking the survey
  self reported, complemented by professional diabetes care provider if possible

CONTACTS AND LOCATIONS:
Overall Officials: Belinda Lennerz, Principal Investigator — Boston Children's Hospital
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified data will be shared with external collaborators.